CLINICAL TRIAL: NCT00306007
Title: Evaluation of the Reliability, Validity, and Acceptability of the London Measure of Unplanned Pregnancy in a U.S. Population of Women
Acronym: LMUP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H1179-27236-01A
Record Dates: First submitted 2006-03-17; First posted 2006-03-22 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Unplanned Pregnancy
Keywords: Pregnancy; Unplanned pregnancy; Psychosocial; Measure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- English prenatal: English speaking women recruited from the general OB/GYN clinic
- Spanish prenatal: Spanish speaking (monolingual) women recruited from the general OB/GYN clinic
- English abortion clinic: English speaking women recruited from the abortion clinic
- Spanish abortion clinic: Spanish speaking (monolingual) women recruited from the abortion clinic

SUMMARY:
The aim of the study is to evaluate the reliability, validity, and acceptability of the London Measure of Unplanned Pregnancy (LMUP) in a U.S. population of women. The researchers hypothesize that the LMUP will be acceptable to a U.S. population and will be reliable and valid.

DETAILED DESCRIPTION:
The concept of "unplanned pregnancy" is used frequently in health research and policy. The majority of tools used to assess unplanned pregnancy planning have not been validated. Recently the London Measure of Unplanned Pregnancy (LMUP) has been developed and validated. The LMUP had been found to be valid and reproducible, but has not been studied outside of the United Kingdom. If we are able to validate this measure in a U.S. population, its use in studies will improve the quality of data about family planning in U.S. women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Basic literacy in English or Spanish needed to participate.

Exclusion Criteria:

* Literacy level lower than 11 years of age

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: target population for this study is pregnant women who present to san Francisco General Hospital (SFGH) Women's Options Center (WOC) for abortion and to the Women's Health Center for prenatal care. The population is racially and ethnically diverse, and the majority are financially challenged and have no insurance or Medicaid.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody Steinauer, MD, MAS, Principal Investigator — University of California, San Francisco; Diane Morof, MD, MSc, Study Director — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States